CLINICAL TRIAL: NCT05080361
Title: Rechallenge of Rapidly Accelerated Fibrosarcoma B-type (BRAF) +/- Mitogen-activated Extracellular Signal-regulated Kinase (MEK) Inhibitors Following an Adverse Event in Patients With Cancer
Brief Title: Rechallenge of BRAF +/- MEK Inhibitors Following an Adverse Event in Patients With Cancer
Acronym: BRAFREC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: BRAFREC
Record Dates: First submitted 2021-04-28; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — MEK inhibitor I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Reports of adverse events associated with the use of BRAF +/- MEK inhibitors: Reports of adverse event (individual case safety reports) from Vigibase, the World Health Organization pharmacovigilance database related to the use of BRAF +/- MEK inhibitors from inception (1986) until March, 1, 2021 will be extracted.
  Cases concurrently reporting on immune checkpoint inhibitor therapies will be excluded.
  Interventions: Drug: BRAF inhibitor

INTERVENTIONS:
Drug: BRAF inhibitor — Reports of adverse events occurring in patients treated with at least one BRAFi or MEKi as reported in the individual case safety reports.
  Other Names: MEK inhibitor

SUMMARY:
Very little data are published on the safety of a rechallenge with a BRAF inhibitor or combination of BRAF and MEK inhibitor (BRAFi and MEKi) after an adverse event (AE). This study aimed at identifying the recurrence rate of the same AE after a BRAFi +/- MEKi rechallenge in patients with cancer and the factors associated to the recurrence.

DETAILED DESCRIPTION:
This is an observational, cross-sectional, pharmacovigilance cohort study. AEs were extracted from safety reports from the World Health Organization database VigiBase®, to evaluate the safety of a rechallenge with a BRAF inhibitor or combination of BRAF and MEK inhibitor (BRAFi and MEKi) after an adverse event (AE) in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive AE cases associated with BRAFi and MEKi therapy. Combination therapy cases, where BRAFi were concurrently reported with MEKi will be identified, as well as the combination therapy regimen (V+C, D+T, E+B). We will not study MEKi monotherapy cases

Exclusion Criteria:

* MEKi monotherapy cases
* Cases concurrently reporting on immune checkpoint inhibitor therapies

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population is made of individual case safety reports from the World Health Organization pharmacovigilance database VigiBase, where patients had an adverse event following BRAF+/-MEKi therapy intakes.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | Up to the date of the individual case safety report notification in VigiBase(r), assessed up to 10 years
  The primary outcome is the rate of recurrence of the same AE after a BRAFi+/- MEKi rechallenge among informative rechallenges The recurrence rate will be obtained by dividing the number of cases with an AE recurrence by the number of informative rechallenges and will be expressed as a percentage

SECONDARY OUTCOMES:
Comparison of rechallenge and non-rechallenge cases | Up to 10 years
  Baseline characteristics (initial adverse event, cancer indication, age, sex) Measurements are the Medical Dictionary for Regulatory Activities preferred terms for adverse events and cancer indications, the Anatomical and Therapeutical Class for drugs. Age is categorized (18-45, 45-64, 65-74, > 75y.o.), sex (male, female).
Factors associated with the recurrence after a rechallenge among informative rechallenges (i.e. variables associated with a higher recurrence rate, in a regression model) | Up to 10 years
  Across baseline characteristics (initial adverse event, cancer indication, age, sex). Measurements are the Medical Dictionary for Regulatory Activities preferred terms for adverse events and cancer indications, the Anatomical and Therapeutical Class for drugs. Age is categorized (18-45, 45-64, 65-74, > 75y.o.), sex (male, female).
  The recurrence is defined as a second occurrence of an initial adverse event after the treatment was reintroduced. It is a dichotomous outcome.
  Data will be analyzed through a regression model, so as to determinate which of these covariates are associated with a higher recurrence rate.
Rate of occurrence of a different AE after a monotherapy or combination therapy rechallenge (among informative rechallenges) | Up to the date of the individual case safety report notification in VigiBase(r), assessed up to 10 years
  The occurrence rate will be obtained by dividing the number of cases with another AE that occurred following a treatment rechallenge by the number of informative rechallenges and will be expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Charles Dolladille, Principal Investigator — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: No
Data for this study are available at http://www.vigiacess.org/. Dissemination to study participants / researchers is not possible outside of the dedicated website.